CLINICAL TRIAL: NCT02654704
Title: Vaccination Responses in Young and Older Adults
Status: Terminated | Type: Observational
Why Stopped: There was insufficient enrollment of subjects.
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, George Mias, Associate Professor, Michigan State University
Other Study IDs: 15-1029F
Record Dates: First submitted 2016-01-10; First posted 2016-01-13 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Individuality; Healthy; Asthma; Immune System and Related Disorders
Keywords: Personalized Medicine; Precision Medicine
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If the volunteers agree,tissue is stored for usage in future research without identifiers. This includes cells from blood and saliva and extracted DNA, RNA and protein. The cells may be used to grow a new cell line that may be maintained in the laboratory.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Healthy Young Adults: Healthy young adults aged 18-25. Vaccination in all cohorts/groups.
  Interventions: Biological: Pneumococcal Vaccination
- Asthma Young Adults: Young adults aged 18-25 with asthma. Vaccination in all cohorts/groups.
  Interventions: Biological: Pneumococcal Vaccination
- Immunocompromised Young Adults: Young adults aged 18-25 that are immunocompromised (e.g. following treatment for leukemia).
  Vaccination in all cohorts/groups.
  Interventions: Biological: Pneumococcal Vaccination
- Healthy Older Adults: Healthy older adults aged 55+ Vaccination in all cohorts/groups.
  Interventions: Biological: Pneumococcal Vaccination
- Asthma Older Adults: Older adults 55+ with asthma. Vaccination in all cohorts/groups.
  Interventions: Biological: Pneumococcal Vaccination
- Immunocompromised Older Adults: Older adults aged 55+ that are immunocompromised (e.g. following treatment for leukemia).
  Vaccination in all cohorts/groups.
  Interventions: Biological: Pneumococcal Vaccination

INTERVENTIONS:
Biological: Pneumococcal Vaccination — The individuals will be followed to observe their immune system activation, following their vaccination with the standard Pneumococcal Polysaccharide Vaccine (PPSV23) as approved by the FDA.

SUMMARY:
To follow longitudinally healthy and immune-compromised responses to pneumococcal vaccination, in 60+ individuals towards the development of personalized medicine implementation (minimum enrollments in 2 age categories: young adults[18-25], older adults [55+], within each category: 10+ healthy, 10+ asthma, 10+ immune-compromised [e.g. leukemia or autoimmune disorders]). The approach will profile thousands of molecular components utilizing high-throughput technologies and integrate these data to obtain personalized immune response to vaccination. The study will provide insights into immune response mechanisms specific to asthmatics, immune compromised and healthy individuals, as well as in response to vaccination. Additionally the differences in dynamic response across the two age groups will be investigated.

DETAILED DESCRIPTION:
The primary investigation involves integrative multi-omics monitoring of individuals following their pneumonia vaccination over twelve time points. Genomic sequencing will be used to evaluate the volunteer's genomic risks based on variants with known disease association. Full transcriptome (via RNA-Sequencing), proteome and metabolome profiling (via mass spectrometry) will be performed per time-point. This will allow the dynamic monitoring of thousands of molecular components and their responses to vaccination, capturing both the initial innate response reaction in addition to the adaptive response and return to baseline. This study involves a simple blood draw, saliva collection, standard FDA-approved pneumococcal vaccine administration and Spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Participants ages 18 to 25 years old, or 55 and older, who have been diagnosed with asthma, other immune-compromising condition (e.g. Leukemia treated, Pulmonary disorders) or are healthy.

Exclusion Criteria:

* Subjects may not participate in this study if any of the following applies:

The potential subjects have already been vaccinated with PPSV23. Subjects have special risks attendant to venipuncture. Existence of any medical conditions that study investigators believe will interfere with the study participation or evaluation of results. This includes subjects on immunosuppressive medications and/or glucocorticoids.

Mental incapacity and/or cognitive impairment that would preclude adequate understanding of, or cooperation with, the study protocol.

For female participants: subjects will be excluded if pregnant. There are no known risks to pregnant women from the PPSV23 vaccine (also indicated in the Vaccine Information Statement (VIS) attachment provided to participants), and there is no additional risk associated with becoming pregnant during the study. However, as pregnancy affects immune system responses, this may affect the molecular readout in this study and introduce confounding factors in the analysis by the investigators. If a participant is already enrolled and becomes pregnant during this study, the investigators will temporarily withdraw them from the study from the day the participants become pregnant. If the participants would like to stay in the study, the investigators may continue their participation after their delivery.

If a participant has any severe allergies (life-threatening) or a participant has ever had a life-threatening allergic reaction after a dose of pneumococcal vaccine, or have a known severe allergy to any part of this vaccine, the participants will be advised not participate.

If a participant is not feeling well on the scheduled day of vaccination, the study coordinators will suggest waiting until the participants feel better. If the participant agrees, the vaccination will be rescheduled for a later date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The initial target enrollment is 60+ individuals in three group classifications [healthy, asthmatic, immune-compromised (e.g. Leukemia patients)], with each group further subdivided into two age groups [Young adults (aged 18-25) or Older adults (aged 55+)], without gender or ethnicity restrictions.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2015-11; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Integrated Omics profile | Through study completion, an average of 2 years
  The study will construct RNA-expression, protein profiles and small molecule profiles on immune cells as these change over time prior to and following immune activation by the vaccine. The collective temporal patterns will be used to classify immune response. The outcome measured is an updated integrative Personal Omics Profile as reported at http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3341616/ . This is observational in nature to assess personalized medicine methodology for following immune response.

CONTACTS AND LOCATIONS:
Overall Officials: George I. Mias, PhD, Principal Investigator — Michigan State University
Locations (1):
- Clinical and Translational Science Institute, East Lansing, Michigan, United States

REFERENCES:
- [Background] Chen R, Mias GI, Li-Pook-Than J, Jiang L, Lam HY, Chen R, Miriami E, Karczewski KJ, Hariharan M, Dewey FE, Cheng Y, Clark MJ, Im H, Habegger L, Balasubramanian S, O'Huallachain M, Dudley JT, Hillenmeyer S, Haraksingh R, Sharon D, Euskirchen G, Lacroute P, Bettinger K, Boyle AP, Kasowski M, Grubert F, Seki S, Garcia M, Whirl-Carrillo M, Gallardo M, Blasco MA, Greenberg PL, Snyder P, Klein TE, Altman RB, Butte AJ, Ashley EA, Gerstein M, Nadeau KC, Tang H, Snyder M. Personal omics profiling reveals dynamic molecular and medical phenotypes. Cell. 2012 Mar 16;148(6):1293-307. doi: 10.1016/j.cell.2012.02.009. PMID 22424236
- [Background] Mias GI, Snyder M. Personal genomes, quantitative dynamic omics and personalized medicine. Quant Biol. 2013 Mar;1(1):71-90. doi: 10.1007/s40484-013-0005-3. PMID 25798291